CLINICAL TRIAL: NCT00769158
Title: Combining Medications for the Treatment of Alcohol Dependence: An Inpatient Preliminary Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bankole Johnson (Other)
Responsible Party: Sponsor-Investigator, Bankole Johnson, Chair of Psychiatry and Neurobehavioral Sciences, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13521
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Alcoholism
Keywords: Alcohol; Alcoholism; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Topiramate; Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate + Naltrexone (Experimental): Combination of Topiramate and Naltrexone
  Interventions: Drug: Topiramate and Naltrexone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Topiramate and Naltrexone — Topiramate 200 mg and Naltrexone 50 mg
  Other Names: Topamax and Revia
  Arms: Topiramate + Naltrexone
Other: Placebo — Placebo Comparator
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
We propose to conduct an inpatient pilot study to test the safety and potential efficacy of topiramate and naltrexone in combination for the treatment of alcoholism.

DETAILED DESCRIPTION:
Eight (n = 8) alcohol-dependent research volunteers, not seeking treatment, will complete a placebo-controlled, within-subject cross-over design in which alcohol-related and control cues are presented as stimuli to induce alcohol-seeking behavior under controlled laboratory conditions after repeated dose (chronic) treatment with double-blind doses of placebo or topiramate + naltrexone.Subjects will reside in an inpatient environment for two separate 9-day blocks interspersed by a 1-week washout period. During separate blocks, topiramate + naltrexone and placebo doses will be administered orally on a twice-daily regimen (08:00 h and 20:00 h) for 8 days.Doses will start the evening of day 1 and the last dose will be given the morning of day 8. No doses will be given the evening of day 8 or the morning of day 9. On Days 7 and 8 of the dosing regimen, subjects will receive alcohol and alcohol-related cues or the corresponding control cues.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-R diagnosis of alcohol dependence.
* Currently drinking.
* Good physical health as determined by a complete physical examination, electrocardiogram within normal limits
* Negative pregnancy test at intake. Women of childbearing potential will be placed on oral contraceptives and also will be expected to use barrier and spermicide as an additional form of contraception if sexually active.
* Literate in English language, and able to read, understand, and complete rating scales and questionnaires accurately.
* Willingness to comply with study procedures and protocol including agreement to overnight stay at the human laboratory. Compliance with the alcohol, tobacco, and drug-free environment regulations at the human laboratory is also a condition of enrollment.
* Written informed consent.

Exclusion Criteria:

* Expression of desire for immediate treatment for alcohol or drug addiction.
* History of mental illness that warrants treatment or would preclude safe participation in the protocol except nicotine dependence, as determined by mental status and psychiatric interview using the Structured Clinical Interview for DSM-IV.
* Acute or chronic organic brain syndrome, schizophrenia, bipolar disorder, or any psychotic disorder.
* Significant medical illness as determined by history and/or complete physical examination.
* Uncontrolled uterine or cervical bleeding.
* History of blood clots.
* Past problems with oral contraceptive pills.
* Gross neurological disease.
* Mental retardation.
* Neurocognitive functioning >1.5 standard deviation below expected range. If neurocognitive functioning test is >1.5 standard deviation below expected range
* Clinically significant abnormalities on the electrocardiogram
* History of ischemic heart disease or myocardial infarction.
* History of glaucoma or uncontrolled symptomatic thyroid disease.
* Current infective hepatitis as evidenced by clinical manifestations. If hepatitis is suspected, a hepatitis antibody/antigen screen will be done.
* Positive pregnancy test.
* Women 35 and above who smoke will be excluded from participating in this research study.
* Participation in a human laboratory or clinical study within the last 30 days.
* Clinically significant laboratory screening test (LST) results on hematology, chemistry, or urine analysis.
* History of any severe or life-threatening reaction to topiramate or naltrexone
* Past or current history of seizures disorder.
* Past or current history of kidney stones.
* Use of any carbonic anhydrase medication.
* Being treated with any medication with potential interactions with alcohol or naltrexone.
* Pending imprisonment.
* For smokers, previous adverse reaction to nicotine patch
* Reporting no experience of craving for alcohol
* Postmenopausal women will not be recruited into this study.
* Chronic use of NSAIDs

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety of this novel combination of topiramate and naltrexone. To evaluate the efficacy of topiramate and naltrexone in combination for the treatment of alcoholism. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, DSc,MD.PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - UVA CARE, Charlottesville, Virginia
  - UVA CARE Richmond, Richmond, Virginia